CLINICAL TRIAL: NCT05383573
Title: Pediatric ANCA Associated-vasculitis : Latest Clinical Review and Therapeutic Outcomes. A Retrospective Epidemiological Study on a French Cohort
Brief Title: Pediatric ANCA Associated-vasculitis
Acronym: PediANCA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8217
Record Dates: First submitted 2022-05-12; First posted 2022-05-20 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: ANCA-Associated Vasculitis
Keywords: ANCA-Associated Vasculitis; Pediatric ANCA; Vasculitis
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Vasculitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The incidence in pediatrics is very low (about 0.5 per million according to a French study) and therefore the data on the pathology very poor, especially on the therapeutic level.

Without appropriate treatment, the mortality rate of the pathology is very high.

Existing treatments are almost exclusively composed of immunomodulatory and/or immunosuppressive treatments.

Complications related to pathology and iatrogeny are among the first causes of mortality from this pathology and deserve to be studied in order to be known and if possible avoided. The purpose of the study is to achieve a national comparison of clinical and therapeutic practices.

ELIGIBILITY:
Inclusion criteria:

* Minor subject (<18 years old)
* Diagnosis of ANCA vasculitis according to the international criteria for defining the pathology, GPA or MPA form between 2011 and 2020.
* Subject (and/or his parental authority) who has not expressed, after being informed, his opposition to the reuse of his data for the purposes of this research.

Exclusion criteria:

* Subject (or his parents) having expressed his (their) opposition to participating in the study
* Patients with vasculitis has ANCA in the form of EGPA
* Associated pathologies that cannot be related to the diagnosis of ANCA vasculitis and whose prognosis can lead to biases in the efficacy and/or complications related to treatments.

Ages: 1 Year to 17 Years | Sex: All
Age Groups: Child
Study Population: Minor subject (<18 years old) with diagnosis of ANCA vasculitis according to the international criteria for defining the pathology, GPA or MPA form between 2011 and 2020.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Retrospective study of clinical and therapeutic practices at the national level. | Files analysed retrospectively from January 01, 2011 to December 31, 2020 will be examined]

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Pédiatrie 1 - CHU de Strasbourg - France, Strasbourg, France